CLINICAL TRIAL: NCT02343523
Title: Pilot Study of the Quanttus Device for Monitoring of Patients With Congestive Heart Failure
Brief Title: Pilot Study of the QI Device for Monitoring of Patients With Congestive Heart Failure
Status: Completed | Type: Observational
Sponsor: Scripps Translational Science Institute (Other)
Responsible Party: Principal Investigator, Steven Steinhubl, Prinicipal Investigator, Scripps Translational Science Institute
Other Study IDs: 14-6510
Record Dates: First submitted 2014-12-18; First posted 2015-01-22 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Heart Failure
Keywords: Wearable device; Wrist-watch; Longitudinal monitoring; Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
The present study proposes to utilize a novel, wearable device, QI Device, which has multiple sensors embedded in a "wrist-watch" in order to explore its monitoring capabilities in individuals with congestive heart failure.

DETAILED DESCRIPTION:
The QI Device is a self-contained, reusable, rechargeable, battery-powered, wrist-watch that simultaneously tracks and records a number of physiological health related parameters such as heart rate, blood pressure, respiratory rate, temperature, and motion/position. One advantage of this device over current home diagnostic systems is the capability for longitudinal monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Adults over age 18
* Own, and comfortable using, a home computer with internet access (Phase 2 only)
* Acute hospitalization with a primary diagnosis of acute decompensated heart failure (ADHF) diagnosed on the basis of all of the following:

  1. Symptoms:

     * Onset or worsening of dyspnea within the past 2 weeks
  2. Physical exam (at least 1 present):

     * Rales/ Crackles on auscultation
     * Elevated JVP > 10 cmH2O
     * Weight gain
     * LE edema
  3. Diagnostic imaging/ labs (at least 1 present):

     * Evidence of pulmonary congestion or edema on chest X-ray/ chest CT
     * Elevated BNP or NT-pro-BNP (age-adjusted)

Exclusion Criteria:

* Psychological or social situation that would make the study difficult for the patient
* Inability to consent
* Chronic atrial fibrillation or other dysrhythmia with a high (>10%) burden of ectopic beats.
* Pregnant women
* Pneumonia - currently, or within the past 30 days
* Non-cardiogenic pulmonary edema (e.g. ARDS)
* Interstitial lung disease
* End-stage renal disease and on Hemodialysis

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population in both phases of the study will be made up of adult men and women admitted to the hospital with a clinical diagnosis of acute decompensated heart failure.
  Phase 1 and Phase 2 will include up to 10 individuals each that meet the following Inclusion criteria and have no Exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2015-01; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
To capture continuous vital signs via a wrist-based wearable physiologic monitor among patients with acute decompensated heart failure (ADHF) in 2 phases | ~7to 30 days
  Phase 1: Will include hospitalized patients admitted to the hospital with a clinical diagnosis of ADHF. Phase 2: Will include patients being discharged from the hospital with a primary clinical diagnosis of ADHF and will be monitored for up to 30 days following hospitalization.

SECONDARY OUTCOMES:
To explore the development of predictive algorithms to allow for the early identification of patients at risk of acute decompensation and/or HF hospitalization. | ~40 days

CONTACTS AND LOCATIONS:
Overall Officials: Steven Steinhuble, MD, Principal Investigator — STSI; Ajay Srivastava, MD, Principal Investigator — STSI
Locations (1):
- Scripps Health, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No